CLINICAL TRIAL: NCT05540938
Title: Reevaluation of Original Research Results of Integrated Traditional Chinese and Western Medicine and Transformation of Hospital Preparations: Post-marketing Re-evaluation of WangBi Granules for Rheumatoid Arthritis
Brief Title: Post-marketing Re-evaluation of WangBi Granules for Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other); The 980th Hospital of PLA Joint Logistics Support Force (Unknown); The Second Affiliated Hospital of Zhejiang Chinese Medical University (Other); Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Zihan Wang, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-NHLHCRF-LX-02-02
Record Dates: First submitted 2022-09-10; First posted 2022-09-15 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): Methotrexate 7.5-15mg qw plus tofacitab 5mg bid, combined with Wangbi granules 12.0g tid, treatment course 3 months.
  Interventions: Drug: Wangbi granules
- control group (Active Comparator): Methotrexate 7.5-15mg qw plus tofacitab 5mg bid, combined with Wangbi granules simulant 12.0g tid, treatment course 3 months.
  Interventions: Drug: Wangbi granules simulant

INTERVENTIONS:
Drug: Wangbi granules — Methotrexate 7.5-15mg qw plus tofacitab 5mg bid, combined with Wangbi granules 12.0g tid, treatment course 3 months.
  Arms: treatment group
Drug: Wangbi granules simulant — Methotrexate 7.5-15mg qw plus tofacitab 5mg bid, combined with Wangbi granules simulant 12.0g tid, treatment course 3 months.
  Arms: control group

SUMMARY:
The group used a randomized controlled trial to conduct a post-marketing re-evaluation study of Wangbi granules. The study was conducted to observe the degree of clinical remission in rheumatoid arthritis patients with low disease activity after standard methotrexate and tofacitinib citrate treatment, using a combination of Chinese and Western medicine treatment with Wangbi granules. The study aims to provide evidence-based medical evidence to improve the clinical efficacy of rheumatoid arthritis, enhance the depth of remission, and improve the diagnosis and treatment of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Meeting the 1987 ACR or 2010 ACR/EULAR diagnostic criteria.
3. Meeting the diagnostic criteria of Chinese medicine for Kidney deficiency and dampness and stasis blocking channels in Chinese medicine.
4. Rheumatoid arthritis disease activity score DAS28 of 2.6 to 3.2.
5. Regularly taking methotrexate 7.5-15 mg qw and tofacitab 5 mg bid before enrollment and stable treatment regimen for more than 4 weeks.
6. Voluntary participation and signed written informed consent.

Exclusion Criteria:

1. Patients taking immunosuppressive drugs other than traditional DMARDs for rheumatoid arthritis within 3 months prior to enrollment (traditional DMARDs include hydroxychloroquine sulfate, methotrexate, salazosulfapyridine tablets, and raglan polysaccharide tablets, among others).
2. Organ transplant recipients, patients with malignant tumors, patients with heart, brain, liver (ALT/AST > 3 times the normal upper limit), kidney (Ccr <60ml/min) and other important organ function impairment or hematological system diseases.
3. Psychiatric disorders such as cognitive disorders, depression, anxiety disorders, somatic dysfunction, cerebral infarction, cerebral hemorrhage, epilepsy, TIA, myelitis, demyelinating lesions and other central neurological disorders, or peripheral neurological disorders such as restless legs syndrome. peripheral neurological disorders such as restless legs syndrome.
4. Women and men who are pregnant or breastfeeding or who are planning a pregnancy within the next 6 months; during the trial or within 1 month of the last dose Women of childbearing age who are unable or unwilling to use adequate contraception, or whose spouse is unwilling to use contraception, within one month of the last dose or within one month of the last dose are unwilling to use contraception.
5. Persons with a BMI greater than 35 (kg/m2), allergic to the test drug, or participating in other clinical trials.
6. Other conditions deemed by the investigator to be inappropriate for trial participation (out-of-town patients unable to be followed up, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
DAS28 | 12 weeks
  Disease mobility score for 28 joints, higher scores indicate higher disease activity

SECONDARY OUTCOMES:
Fatigue Scale-14 | 12 weeks
  assessing the patient's fatigue level, the higher the score, the more severe the fatigue
visual analogue scale | 12 weeks
  Patients score according to the level of pain they feel, there are 10 scales from 0-10, with 0 representing no pain and 10 representing severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Wang Z, Lan T, Zhang L, Li Z, Wang X, Zou Q, Wang Y, Li Y, Luo R, Zhang N, Xu Y, Li M, Tao Q. Wangbi granule as a combination therapy to achieve clinical deep remission in rheumatoid arthritis: protocol for a multicenter, triple-blind, randomised, placebo-controlled trial. Chin Med. 2023 Feb 28;18(1):22. doi: 10.1186/s13020-023-00728-6. PMID 36855169